CLINICAL TRIAL: NCT05388786
Title: Complications and Adverse Events in Lymphadenectomy in the Inguinal Area: Delphi Consensus on Adverse Events Definition and Management
Brief Title: Complications and Adverse Events in Lymphadenectomy in the Inguinal Area
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Rene Sotelo, Professor of Clinical Urology, University of Southern California
Other Study IDs: UP-22-00368
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Consensus Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delphi Panel: A team of experts in open inguinal lymphadenectomy, video endoscopic inguinal lymphadenectomy (VEIL), and robotic-assisted video endoscopic inguinal lymphadenectomy (R-VEIL) in the fields of General Surgery, Gynecology Oncology, Surgical Oncology, and Urology will be invited to participate. These experts are identified according to surgical experience, research, and academic interest.
  Interventions: Behavioral: Delphi Questionnaire

INTERVENTIONS:
Behavioral: Delphi Questionnaire — An invitation email, including a link to the survey, will be sent to the panel of experts in ILND for penile cancer, vulvar cancer, and melanoma.
  The Delphi questionnaire will be administered via Welphi.com. In the first survey, panel members will outline the ILND complications and adverse events definition and classification with a series of 5-point Likert scale assessments and options for free-text responses relating to the surgeon's perception.
  The experts will fill out the online questionnaire. For the questions that do not reach a consensus of more than 80% in the first round or need further explanation, additional rounds of the survey may be performed.

SUMMARY:
The investigators aim to create an effective and accurate method to report, define, and classify complications and adverse events during and after Inguinal lymph node dissection (ILND) as part of the staging and treatment for penile cancer, vulvar cancer, and melanoma. In turn, this will become an objective, efficient, and reproducible tool to facilitate comparisons across surgical approaches, techniques, and surgeons.

DETAILED DESCRIPTION:
Inguinal lymph node dissection (ILND) has shown to be a necessary surgery from the oncology standpoint being extensively used as part of the staging process in malignancies of the penis, vulva, or melanoma. Moreover, the ILND has been shown to improve survival if performed in a timely manner. Yet, ILND is linked to a high rate of complications and adverse events.

Complications and adverse events' incidence are frequently used as surrogate markers of quality in surgery. However, there is tremendous heterogeneity in the report in such specifically for this procedure. Even though different classification and grading systems on surgical complications are available. There is a lack of standardization regarding the definition and classification to report ILND complications and adverse events leading to discrepancies across the literature, often interfering with the interpretation of surgical performance and quality.

This study will provide a systematic definition and classification of ILND complications and adverse events, ultimately improving the reporting of such conditions for future studies.

To create an effective and accurate method to report, define, and classify complications and adverse events during and after ILND as part of the staging and treatment for penile cancer, vulvar cancer, and melanoma. In turn, this will become an objective, efficient, and reproducible tool to facilitate comparisons across surgical approaches, techniques, and surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Experts in open inguinal lymphadenectomy
* Experts in video endoscopic inguinal lymphadenectomy (VEIL)
* Experts in robotic video endoscopic inguinal lymphadenectomy (R-VEIL)
* Authors with at least one publication in ILND for penile cancer, vulvar cancer, or melanoma

Exclusion Criteria:

* Panelists who were not able to commit to all rounds of the modified Delphi process will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A team of experts in open inguinal lymphadenectomy, video endoscopic inguinal lymphadenectomy (VEIL), and robotic-assisted video endoscopic inguinal lymphadenectomy (R-VEIL) in the fields of General Surgery, Gynecology Oncology, Surgical Oncology, and Urology will be invited to participate. These experts are identified according to surgical experience, research, and academic interest.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Degree of consensus | 1 month
  The level of agreement for all statements achieving consensus from the expert panel; consensus is predefined as ≥ 80% of the panel rating a given statement

CONTACTS AND LOCATIONS:
Overall Officials: Rene Sotelo, MD, Principal Investigator — University of Southern California; Giovanni Cacciamani, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chipollini J, Tang DH, Gilbert SM, Poch MA, Pow-Sang JM, Sexton WJ, Spiess PE. Delay to Inguinal Lymph Node Dissection Greater than 3 Months Predicts Poorer Recurrence-Free Survival for Patients with Penile Cancer. J Urol. 2017 Dec;198(6):1346-1352. doi: 10.1016/j.juro.2017.06.076. Epub 2017 Jun 23. PMID 28652123
- [Background] Gkegkes ID, Minis EE, Iavazzo C. Robotic-assisted inguinal lymphadenectomy: a systematic review. J Robot Surg. 2019 Feb;13(1):1-8. doi: 10.1007/s11701-018-0823-4. Epub 2018 May 5. PMID 29730734
- [Background] Munoz Guillermo V, Rosino Sanchez A, Rivero Guerra A, Barcelo Bayonas I, Pardo Martinez A, Jimenez Peralta D, Carrillo George C, Pietricica BN, Izquierdo Morejon E, Cruces de Abia FI, Romero Hoyuela A, Hita Villaplana G, Fernandez Aparicio T. [Video endoscopic inguinal lymphadenectomy in penile cancer: Systematic review.]. Arch Esp Urol. 2019 Dec;72(10):992-999. Spanish. PMID 31823847
- [Background] Mitropoulos D, Artibani W, Graefen M, Remzi M, Roupret M, Truss M; European Association of Urology Guidelines Panel. Reporting and grading of complications after urologic surgical procedures: an ad hoc EAU guidelines panel assessment and recommendations. Eur Urol. 2012 Feb;61(2):341-9. doi: 10.1016/j.eururo.2011.10.033. Epub 2011 Oct 29. PMID 22074761
- [Background] Dindo D, Clavien PA. What is a surgical complication? World J Surg. 2008 Jun;32(6):939-41. doi: 10.1007/s00268-008-9584-y. No abstract available. PMID 18414942
- [Result] Nabavizadeh R, Petrinec B, Necchi A, Tsaur I, Albersen M, Master V. Utility of Minimally Invasive Technology for Inguinal Lymph Node Dissection in Penile Cancer. J Clin Med. 2020 Aug 3;9(8):2501. doi: 10.3390/jcm9082501. PMID 32756502